CLINICAL TRIAL: NCT00186017
Title: Double-Blind Placebo-Controlled Olanzapine Add-on Therapy in the Treatment of Acute Syndromal and Subsyndromal Exacerbations in Bipolar Disorders
Brief Title: Short Term Rescue Study of Olanzapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Terrence Ketter, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 79897; F1D-US-X279 (Other Grant/Funding Number: Eli Lilly)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine/Zyprexa (Experimental): Olanzapine/Zyprexa 2.5 mg up to 8 per day for 1 week
  Interventions: Drug: Olanzapine/Zyprexa
- Placebo (Placebo Comparator): Placebo was taken in the same manner as olanzapine with up to 8 per day for 1 week
  Interventions: Drug: Olanzapine/Zyprexa

INTERVENTIONS:
Drug: Olanzapine/Zyprexa — Olanzapine was started at 2.5-10mg/day and adjusted by 2.5-5mg/day on a daily basis with a maximum dose of 20mg/day.
  Other Names: Zyprexa

SUMMARY:
We will assess the effect of olanzapine compared to placebo added to prior treatment on CGI-S in a one-week randomized double-blind study. We will also assess the effect of olanzapine added to prior treatment on CGI-S in an eight-week open treatment study. In addition, we will assess the effect of olanzapine on Young Mania Rating Scale (YMRS), Hamilton and Montgomery-Asberg Depression Rating Scales (HDRS, and MADRS), and Hamilton Anxiety Rating Scales (HARS) in the above paradigms. We will also assess the influence of presentation severity (CGI-S) and polarity (mood elevation versus depression) on olanzapine response. Finally, we will assess safety and tolerability of olanzapine in the above paradigms.

We hypothesize that in diverse mild syndromal and subsyndromal exacerbations of BD in outpatients, randomized double-blind flexibly dosed olanzapine added to prior treatment (including no treatment) will yield greater CGI-S improvement than placebo by the end of one week, and that such improvement will persist over one week of open continuation treatment.

DETAILED DESCRIPTION:
Development and marketing of new therapies for bipolar disorders (BD) has typically entailed performing double-blind placebo-controlled trials in acute mania maintenance studies and more recently acute depression studies. Such an approach addresses BD primarily in terms of episodes and has the strength of studying levels of pathology sufficiently high to permit detection of treatment effects, and guiding clinicians when they encounter syndromal mood episodes. However, this approach has the important limitation of not addressing an important unmet clinical need, namely the management of subsyndromal symptoms. Indeed, emerging data suggest that in BD subsyndromal symptoms compared to syndromal episodes are far more pervasive. Also such an approach runs the risk of not paying sufficient attention to the disorder construct, in a sense permitting preoccupation with syndromal episodes to carry more importance than the disorder.

We will assess the effect of olanzapine compared to placebo added to prior treatment on CGI-S in a one-week randomized double-blind study. We will also assess the effect of olanzapine added to prior treatment on CGI-S in an eight-week open treatment study. In addition, we will assess the effect of olanzapine on Young Mania Rating Scale (YMRS), Hamilton and Montgomery-Asberg Depression Rating Scales (HDRS, and MADRS), and Hamilton Anxiety Rating Scales (HARS) in the above paradigms. We will also assess the influence of presentation severity (CGI-S) and polarity (mood elevation versus depression) on olanzapine response. Finally, we will assess safety and tolerability of olanzapine in the above paradigms.

ELIGIBILITY:
Inclusion Criteria:Patients must meet the following criteria to be eligible to participate in the study:

* Male or female outpatients, 18 to 70 years of age
* Female patients of childbearing potential must be using a medically accepted means of contraception
* Able to communicate intelligently with the investigator, and study coordinator
* Able to give informed consent
* DSM-IV diagnosis of bipolar I, bipolar II, cyclothymic disorder or bipolar disorder not otherwise specified, experiencing an acute exacerbation of their illness at Visit 1 (hypomania, subsyndromal depression, hypomania and subsyndromal depression, depression and hypomania, or depression if diagnosed with bipolar II) as verified by SCID-I/P
* CGI-BP Overall Severity score greater than or equal to mildly ill at Visit 1
* Must have been on prior medications for at least 2 weeks (6 weeks for fluoxetine) immediately prior to study entry Exclusion Criteria:Patients may not participate in the study if they have any of the following conditions:
* Pregnant, nursing, or intending to become pregnant during the study
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease such that hospitalization for the disease is anticipated within 3 months or death is anticipated within 3 years.
* A history of seizure disorder
* History of leukopenia without a clear and resolved etiology.
* DSM-IV substance (except nicotine or caffeine) dependence within the past month
* Judged clinically to be at serious suicidal risk
* Participation in clinical trial of another investigational drug within 1 month (30 days) prior to study entry.
* Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to study entry
* Treatment resistance, non-response, or intolerability with olanzapine by the investigator's judgment
* Treatment with clozapine within 3 months prior to study entry
* Treatment with remoxipride within 6 months (180 days) prior to study entry
* Treatment with an oral antipsychotic within 2 days prior to study entry
* A course of ECT (electroconvulsive therapy) in the preceding 4 weeks
* Excluded mood symptoms noted in Table 1 [of protocol]
* Unstable thyroid pathology and treatment-initiated or altered within the past 3 months
* Meet criteria for antisocial personality disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Arthur Ketter, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford University Bipolar Disorders Clinic — http://bipolar.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine/Zyprexa: Olanzapine/Zyprexa 2.5 mg up to 8 per day for 1 week
  Olanzapine/Zyprexa
- Placebo: Placebo
  Olanzapine/Zyprexa
Period: Overall Study
Arm/Group | Olanzapine/Zyprexa | Placebo
Started | 25 | 25
Completed | 23 | 22
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine/Zyprexa | Placebo | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12) | 42.9 (9.9) | 40.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 17 | 13 | 30
  Race/Ethnicity: Non-White | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45
Bipolar Subtype [Number; unit: participants]
  Bipolar 1 | 12 | 11 | 23
  Bipolar 2 | 11 | 7 | 18
  Bipolar NOS | 0 | 4 | 4
CGI-BP_OS [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions-Bipolar Version-Overall Severity of Illness (CGI-BP-OS) Scale is 0-7 0=not Assessed
  1=Normal 7=Worst
  units on a scale | 4.8 (.8) | 4.7 (.8) | 4.8 (.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in CGI-BP-OS After 1 Week of Treatment
Description: The Clinical Global Impression - bipolar version - overall severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not ill; 2, minimally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, very severely ill
Time Frame: Baseline, 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo up to 8 per day for 1 week
Arm/Group | Olanzapine/Zyprexa | Placebo
Number analyzed (Participants) | 23 | 22
units on a scale | -1.4 (0.9) | .8 (1.1)
Statistical Analysis 1: Comparison: Olanzapine/Zyprexa vs Placebo; Test type: Superiority or Other; p = .08, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Mean Change in YMRS After 1 Week of Treatment
Description: The Young Mania Rating Scale (YMRS) scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. Responses to each item are summed with a higher score indicating more mania symptoms endorsed.
  Scale:0-60 0=Good 60=Bad
Time Frame: Baseline, 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo
Arm/Group | Olanzapine/Zyprexa | Placebo
Number analyzed (Participants) | 23 | 22
units on a scale | -6.0 (6.7) | -3.3 (4)
Statistical Analysis 1: Comparison: Olanzapine/Zyprexa vs Placebo; Test type: Superiority or Other; p > .1, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mean Change in MADRS After 1 Week of Treatment.
Description: Montgomery-Asberg Depression Rating Scales (MADRS) is a multi-item clinician tool assessing depression. Each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Higher MADRS score indicates more severe depression.
Time Frame: Baseline, 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine/Zyprexa | Placebo
Number analyzed (Participants) | 23 | 22
units on a scale | -12.3 (9.5) | -6.8 (10.5)
Statistical Analysis 1: Comparison: Olanzapine/Zyprexa vs Placebo; Test type: Superiority or Other; p > .1, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mean Change in Hamilton Anxiety Rating Scales (HAM-A)
Description: The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms, and is still widely used today in both clinical and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The HAM-A does not provide any standardized probe questions. Despite this,the reported levels of interrater reliability for the scale appear to be acceptable.
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Baseline, 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine/Zyprexa | Placebo
Number analyzed (Participants) | 23 | 22
units on a scale | -7.9 (6.3) | -3.8 (6.1)

ADVERSE EVENTS:
Description: Adverse events were systematically collected using a standardized clinical monitoring and treatment form
Groups:
- Placebo: Placebo taken in same manner as study drug up to 8 per day for 1 week
Arm/Group | Olanzapine/Zyprexa | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 22/23 | 20/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olanzapine/Zyprexa (N=23) | Placebo (N=22)
Increased appetite (Gastrointestinal disorders) | 12 | 5
Tremor (Nervous system disorders) | 11 | 2
Sedation (Nervous system disorders) | 14 | 13
Dry mouth (Gastrointestinal disorders) | 18 | 10
Constipation (Gastrointestinal disorders) | 7 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 3
Headache (Nervous system disorders) | 12 | 7
Poor memory (Nervous system disorders) | 14 | 11
Sexual dysfunction (Psychiatric disorders) | 4 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Cramps (Nervous system disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small Sample Size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No